CLINICAL TRIAL: NCT05015348
Title: Effects of Omega-3 Polyenoic Acid on Blood Lipid, Inflammatory Factors and Body Composition in Patients with Hyperlipidemia
Brief Title: Effects of Omega-3 PUFA on Lipids, Inflammatory Factors and Body Composition in Patients with Hyperlipidemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-2908
Record Dates: First submitted 2021-07-24; First posted 2021-08-20 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- O3A arm (Experimental): participants of this arm will be provided with omega-3 PUFA
  Interventions: Other: fish oil with omega-3 PUFA
- placebo arm (Placebo Comparator): participants of this arm will be provided with same amount of corn oil as placebo
  Interventions: Other: placebo

INTERVENTIONS:
Other: fish oil with omega-3 PUFA — 3.6g per day fish oil with omega-3 PUFA (EPA+DHA)
  Arms: O3A arm
Other: placebo — palm oil as placebo
  Arms: placebo arm

SUMMARY:
Patients with hyperlipidemia will be allocated into intervention or control group randomly. Participants of intervention group will be provided with Omega-3 PUFA, while participants of control group will be provided with placebo which looked same as the drug of intervention group. During the study, all participants can have nutritional counseling and education for low-fat diet. The lipids, inflammatory factors, weight, and body composition will be assessed and recorded before, at the middle, and end of the study.

DETAILED DESCRIPTION:
Randomization tables were generated by the statistician and provided to the investigational pharmacist who distributed the blinded pills to participants.

Participants of intervention group will be provided with Omega-3 PUFA, while participants of control group will be provided with placebo which looked same as the drug of intervention group. During the study, all participants can have nutritional counseling and education for low-fat diet. The lipids, inflammatory factors, weight, and body composition will be assessed and recorded before, at the middle, and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* [1] Gender and age: male or female, 18 years old and above.
* [2] Patients were diagnosed with hyperlipidemia. According to the definition of 2016 guidelines for the prevention and treatment of dyslipidemia in Chinese adults, it meets the clinical diagnostic criteria of hyperlipidemia: hypertriglyceridemia [TG≥1.7mmol/L]; Or mixed with TC≥5.2mmol/L]; Or mixed with LDL-C≥3.4mmol/L].
* [3] Before the study, the subjects fully understood and voluntarily signed the informed consent form, and fully understood the research content, process and possible adverse reactions.
* [4] Those who can eat orally.
* [5] Be able to complete the research according to the requirements of the research protocol and obey the arrangements of doctors and researchers.

Exclusion Criteria:

* [1] Those who are receiving lipid-lowering drugs.
* [2] Hyperlipidemia caused by secondary causes, such as nephrotic syndrome, hypothyroidism, renal failure, liver disease, systemic lupus erythematosus, glycogen accumulation, myeloma, fat atrophy, acute porphyria, polycystic ovary syndrome, etc; Use diuretics, non cardiac selective β Receptor blockers and glucocorticoids which may cause secondary dyslipidemia.
* [3] Patients with severe internal and external diseases, such as heart, liver and kidney dysfunction, acute myocardial infarction, stroke, intracerebral hemorrhage, acute attack of COPD, respiratory failure, etc. in recent 3 months, patients who have undergone surgery in recent 3 months, or any person who is not suitable to participate in this study after clinician evaluation.
* [4] Have hemorrhagic disease or bleeding tendency.
* [5] Those who have a history of allergy to omega-3 polyenoic acid preparation.
* [6] Pregnant and lactating women.
* [7] Poor compliance, unable to follow up on time or unable to complete the follow-up of medication.
* [8] In the course of diagnosis and treatment, if there is any seriously abnormal metabolism or further intervention is needed, or the patient is no longer suitable for continuing the study through the assessment of the competent physician, he can withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
triglyceride | 3 months
  triglyceride in mmol/L
cholesterol | 3 months
  cholesterol in mmol/L
LDL-C | 3 months
  LDL-C in mmol/L
TNF-α | 3 months
  TNF-α in ng/ml
hsCRP | 3 months
  hsCRP in mmol/L
interlukin-6 | 3 months
  IL-6 in ng/ml
body weight | 3 months
  weight in kilogram
BMI | 3 months
  BMI in kg/m2

SECONDARY OUTCOMES:
adiponectin | 3 months
  adiponectin in μg/mL
leptin | 3 months
  leptin in μg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, master, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospita, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No